CLINICAL TRIAL: NCT04258189
Title: A Phase 1, Randomized, Open-label, 4-Period Crossover Study in Healthy Subjects to Assess the Food Effect on a Single Dose of JNJ-64417184 Administered as an Oral Solution
Brief Title: A Study of JNJ-64417184, Administered as an Oral Solution, in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108752; 2019-004189-16 (EudraCT Number); 64417184RSV1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Panel 1: Treatment Sequence ABDC (Experimental): Participants will receive Treatment A (a single dose of JNJ-64417184 [oral solution with preservatives] in fasted condition) in treatment Period 1; followed by Treatment B (a single dose of JNJ-64417184 [oral solution with preservatives] in fed [high-fat meal] condition) in treatment Period 2; followed by Treatment D (a single dose of JNJ-64417184 [oral solution without preservatives] in fed [high-fat meal] condition) in treatment Period 3, followed by Treatment C (a single dose of JNJ-64417184 [oral solution without preservatives] in fasted condition) in treatment Period 4 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Panel 1: Treatment Sequence BCAD (Experimental): Participants will receive Treatment B in treatment Period 1; followed by Treatment C in treatment Period 2; followed by Treatment A in treatment Period 3, followed by Treatment D in treatment Period 4 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Panel 1: Treatment Sequence CDBA (Experimental): Participants will receive Treatment C in treatment Period 1; followed by Treatment D in treatment Period 2; followed by Treatment B in treatment Period 3, followed by Treatment A in treatment Period 4 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Panel 1: Treatment Sequence DACB (Experimental): Participants will receive Treatment D in treatment Period 1; followed by Treatment A in treatment Period 2; followed by Treatment C in treatment Period 3, followed by Treatment B in treatment Period 4 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Optional Panel 2: Treatment Sequence EFG (Experimental): Participants will receive Treatment E (a single dose of JNJ-64417184 [oral solution with or without preservatives] in fasted condition) in treatment Period 1; followed by Treatment F (a single dose of JNJ-64417184 [oral solution with or without preservatives] in fed [high-fat meal] condition) in treatment Period 2; followed by Treatment G (a single dose of JNJ-64417184 [oral solution with or without preservatives] in fed [high-fat meal] condition) in treatment Period 3 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Optional Panel 2: Treatment Sequence FGE (Experimental): Participants will receive Treatment F in treatment Period 1; followed by Treatment G in treatment Period 2; followed by Treatment E in treatment Period 3 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Optional Panel 2: Treatment Sequence GEF (Experimental): Participants will receive Treatment G in treatment Period 1; followed by Treatment E in treatment Period 2; followed by Treatment F in treatment Period 3 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Optional Panel 2: Treatment Sequence GFE (Experimental): Participants will receive Treatment G in treatment Period 1; followed by Treatment F in treatment Period 2; followed by Treatment E in treatment Period 3 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Optional Panel 2: Treatment Sequence EGF (Experimental): Participants will receive Treatment E in treatment Period 1; followed by Treatment G in treatment Period 2; followed by Treatment F in treatment Period 3 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184
- Optional Panel 2: Treatment Sequence FEG (Experimental): Participants will receive Treatment F in treatment Period 1; followed by Treatment E in treatment Period 2; followed by Treatment G in treatment Period 3 on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each study drug intakes.
  Interventions: Drug: JNJ-64417184

INTERVENTIONS:
Drug: JNJ-64417184 — Single dose of JNJ-64417184 solution (with or without preservatives) will be administered orally.

SUMMARY:
The purpose of this study is to assess the food effect on the single-dose pharmacokinetic (PK) of the JNJ-64417184 oral solution, administered as 2 different formulations, in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI; weight [kg]/height^2 [m^2]) between 18.0 and 30.0 kilogram per meter square (kg/m^2), extremes included, and a body weight not less than 50.0 kg at screening
* Healthy on the basis of physical examination, medical and surgical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study
* Healthy on the basis of clinical laboratory tests performed at screening
* Must have a normal 12-lead electrocardiogram (ECG) (triplicate) at screening
* Female participant must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta- hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1

Exclusion Criteria:

* History of liver or renal dysfunction significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Past history of cardiac arrhythmias (example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Any evidence of heart block or bundle branch block at screening
* Current human immunodeficiency virus type-1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* A history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-64417184 | Up to Day 6
  Cmax is the maximum observed plasma analyte concentration.
Area Under the Concentration-time Curve from Time Zero to the Last Measurable Concentration (AUC [0-last]) of JNJ-64417184 | Up to Day 6
  AUC (0-last) is area under the plasma analyte concentration-time curve (AUC) from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ-64417184 | Up to Day 6
  AUC (0-infinity) is the area under the plasma analyte concentration-time curve (AUC) from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) analyte concentration; and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 28 days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment.
Acceptability of the JNJ-64417184 Formulation as Assessed by Participant | Up to 28 days
  The acceptability of the JNJ-64417184 formulations will be assessed by the participants using a questionnaire designed to rate the taste and smell as well as the overall acceptability of the formulations. The questionnaire will consist of a visual analogue scale to rate 5 items (sweetness, bitterness, aroma type, aroma strength, and smell) as well as overall acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency